CLINICAL TRIAL: NCT01992042
Title: Novel Window of Opportunity Trial to Evaluate the Impact of Statins to Oppose Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIN-STOPCa_001
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fluvastatin; pimonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluvastatin/Pimonidazole (Experimental): Patients will take 40mg BID of fluvastatin. The day before surgery patients will take a single dose of pimonidazole that will be calculate based on body surface area.
  Interventions: Drug: Fluvastatin; Drug: Pimonidazole

INTERVENTIONS:
Drug: Fluvastatin — HMG-CoA reductase inhibitors that lowers cholesterol levels. 40mg twice daily
  Other Names: Lescol
Drug: Pimonidazole

SUMMARY:
This research study provides a novel opportunity to examine the intra-prostatic tumour inhibitory effects of statins in men with prostate cancer undergoing surgery.

ELIGIBILITY:
The study population will consist of patients with localized prostate cancer that have elected radical prostatectomy as a primary treatment. Eligible patients will have prostate cancer that is Gleason Score ≥ 7.

Patients who meet all of the following inclusion criteria will be eligible to participate in this study:

1. Men >18 and < 75 years of age
2. Willing and able to provide informed consent, either alone or with the aid of a translator
3. Histologically confirmed prostate cancer as determined by transrectal ultrasound (TRUS) guided prostate biopsy performed within 6 months of study enrolment
4. Prostate cancer that is Gleason grade ≥ 7 involving at least 30% of one unfragmented biopsy core
5. Candidates for radical prostatectomy considered surgically resectable, either open or robotic, by urologic evaluation
6. Normal organ and marrow function as defined by the following criteria:

   i. absolute neutrophil count >1,500/uL

   ii. platelets >100,000/uL

   iii. total bilirubin <1.5 X institutional ULN

   iv. AST (SGOT) or ALT (SGPT) <1.5 X institutional ULN

   v. creatinine <1.5 X institutional ULN
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1

Exclusion Criteria

Any patient meeting one or more of the following exclusion criteria may not be entered into the study:

1. Previous or current use of neo-adjuvant or hormonal management of prostate cancer (surgical castration or other hormonal manipulation, including GnRH receptor agonists, GnRH receptor antagonists, anti-androgens, estrogens, megestrol acetate and ketoconazole)
2. History of receiving radiation to the pelvic area
3. Past or current use of 5-alpha reductase inhibitors finasteride and/or dutasteride
4. History of bilateral orchiectomy, adrenalectomy, or hypophysectomy
5. Statin use within 2 years of prostate cancer diagnosis
6. Known hypersensitivity towards any component of the investigational medicinal product.
7. Previous history or presence of another malignancy, other than prostate cancer or treated squamous / basal cell carcinoma of the skin, within the last five years
8. Clinically significant laboratory abnormalities (e.g. severe renal or hepatic impairment) which in the judgment of the Investigator would affect the patient's health or the outcome of the trial
9. Clinically significant disorder (other than prostate cancer) including, but not limited to, renal, haematological, gastrointestinal, endocrine, cardiac, neurological, or psychiatric disease, and alcohol or drug abuse or any other condition, which may affect the patient's health or the outcome of the trial as judged by the Investigator
10. Use of natural medicines thought to have endocrine effects on prostate cancer (e.g. saw palmetto and St. John's Wort) 4 weeks prior to enrollment.
11. Use of any drug listed in Prohibited Medications List
12. Mental incapacity or language barrier precluding adequate understanding or co operation
13. Use of an investigational drug within the last 28 days preceding the Screening Visit or longer if considered to possibly influence the outcome of the current trial
14. Patients who are unable or unwilling to undergo MRI testing

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pre and post treatment effect on the Ki-67 proliferation index | Week 8

SECONDARY OUTCOMES:
Comparison of immunohistochemical staining in Biopsy and post-RP tissues | Week 8
  Will measure:
  i. Apoptosis (caspase 3) ii. Signaling (Rap1A, Rap, RhoB) iii. Mevalonate pathway proteins (HMG-CoA reductase, HMG-CoA synthase, SREBP1/2, mevalonate decarboxylase, GGPS1, GGT, FT) iv. Tumour Infiltrating Lymphocytes (TILs), CD3 (T-cells), CD20 (B-cells), CD68 (macrophages), CD56 (NK cells), IDO (negative control)) v. Growth and survival signaling (AKT, P-AKT, ERK, P-ERK)

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network- The Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Longo J, Hamilton RJ, Masoomian M, Khurram N, Branchard E, Mullen PJ, Elbaz M, Hersey K, Chadwick D, Ghai S, Andrews DW, Chen EX, van der Kwast TH, Fleshner NE, Penn LZ. A pilot window-of-opportunity study of preoperative fluvastatin in localized prostate cancer. Prostate Cancer Prostatic Dis. 2020 Dec;23(4):630-637. doi: 10.1038/s41391-020-0221-7. Epub 2020 Mar 13. PMID 32203069